CLINICAL TRIAL: NCT05140473
Title: Identification of the Determinants of the Perceived Workload of Intensive Care and Pediatric Continuous Monitoring Nurses
Brief Title: Identification of the Determinants of the Perceived Workload of Nurses
Acronym: CHARMIREA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211025; 2021-A01542-39 (Other: ID-RCB)
Record Dates: First submitted 2021-11-02; First posted 2021-12-01 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Nurses's Workload
Keywords: Nurses; Workload; Intensive car unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: perceived workload — Perceived workload takes into account the acts and care performed but also the pressure felt of having been efficient in its task, the efforts made and the level of frustration felt.

SUMMARY:
The purpose of this study is to identify the determinants of the perceived workload of intensive care and pediatric continuous monitoring nurses (factors liked to the care service, staff, patients treated)

DETAILED DESCRIPTION:
In intensive care and pediatric continuous monitoring unit (RSCP), the workload of nurses (registered nurses) is high. It is important to distribute the workload correctly among caregivers in order to guarantee the quality and safety of care.

Workload can be measured by different means. The measure of the perceived workload has the advantage of taking into account not only the acts and care performed, but also the time pressure felt, the feeling of having been efficient in its task, the efforts made and the level of frustration felt.

Measuring the workload of RSCP registered nurses will help highlight the factors that may influence the workload. The aim is to allow an adequate distribution of patients between nurses, taking into account the determinants identified during this study.

Primary objective : Measure RSCP's nurses workload

Secondary objectives: Highlight the determinants of the overall perceived workload of RSCP nurses (organizational characteristics, of the individual, of the patient and of his entourage).

Highlight the determinants of each dimension of the perceived workload of RSCP nurses.

The calendar of data collection days will be defined by drawing lots. The day drawn for data collection will proceed normally, with no change in practice for nurses. A study investigator will inform the legal representative (s) of the possible data collection in their child that day and will trace their non-opposition in the medical file.

At the end of the day, registered nurses should collect data relating to family circles and individual characteristics. In addition, nurses must complete a NASA TLX grid for each patient treated during their working time. The grids will be assembled at the end of the day (around 7 p.m.) and handed over to an investigator. The same procedure will apply to the night shift, the grids will be handed over at 7 a.m. to an investigator.

In the following days, the principal investigator will collect the data related to the organizational characteristics and characteristics of the patients.

The perceived workload of nurses working in Intensive care and Continuous Monitoring Unit will be measured for each nurse who has at least 1 patient in charge during a period of 24 hours over 2 days (a day service and a night service, i.e. from 7 a.m. to 7 a.m. / D + 1 ), once a month for a year.

The measurement periods will be drawn at the rate of a period of 24 hours per month for one year, ie 12 periods in total.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses from Pediatric Intensive care and Continuous Monitoring Unit agreeing to participate in the study,
* Having at least one patient in charge over the period considered
* Child regardless of age hospitalized in the Pediatric Intensive care and Continuous Monitoring unit.
* Non-opposition of the legal representative (s) to the collection of data

Exclusion Criteria:

* Nurse in job adaptation training
* Interim nurse
* Nurse not usually working in intensive care
* Reference nurses of the service
* Legal guardian of the child who doesn't speak or understand French

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses works in Pediatric Intensive care and Continuous Monitoring Unit of the Necker Hospital, AP-HP, Paris Child hospitalized in the Intensive care and Continuous Monitoring Unit of the Necker Hospital, AP-HP, Paris
Sampling Method: Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Task Load indeX scale (TLX scale) | 1 day
  TLX scale is a workload scale according to 6 dimensions: mental demands, physical demands, time pressure, performance, effort and frustration.Each dimension is evaluated on a 100-points scale. A total score from 0 to 600 points is obtained. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Seniority in the profession | 1 day
  Seniority in the profession in years Seniority in the service in years Age Previous patient management (at least once in the previous 12 months) Supervision of a student Tutoring a new nurse
Seniority in the service | 1 day
  Seniority in the service in years Seniority in the service in years Age Previous patient management (at least once in the previous 12 months) Supervision of a student Tutoring a new nurse
Age of nurse | 1 day
  Age of nurse in years Day / night work Number of patient transportations Reception of an incoming patient Participation in an ethics meeting
Age of nurse | 1 day
  Age of nurse in years
Previous patient management | 1 day
  Previous patient management (at least once in the previous 12 months)
Supervision of a student | 1 day
  Supervision of a student (yes/no)
Tutoring a new nurse | 1 day
  Tutoring a new nurse (yes/no)
Ratio patient/nurse | 1 day
  Number of patient split by the number of nurse
Period of work | 1 day
  Day / night work
Patient transport | 1 day
  Number of patient transportations outside the ward.
New patient | 1 day
  Reception of an incoming patient
Ethics meeting | 1 day
  Participation of nurse to an ethics meeting
Age of patient | 1 day
  Age of patient in years
Weight of patient | 1 day
  Weight of patient in kilograms
Lengh of Hospitalisation | 1 day
  Number of days in hospital
Glasgow score | 1 day
  Glasgow score of patient. Scored on a total score from 3 to 15 points is obtained. A higher score means a better outcome.
Vascular supply | 1 day
  Type of vascular catheter present on the patient
Supportive system | 1 day
  Number of supportive systems necessary
Treatment | 1 day
  Number of treatments administered / 24 hours
Resuscitation maneuver | 1 day
  Resuscitation maneuver necessary (yes/no)
Death | 1 day
  Death of patient (yes/no)
Family support | 1 day
  Number of hours of presence of at least one of the two parents
Phone calls | 1 day
  Number of phone calls from parents
Family interview | 1 day
  Family interview realised ( Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie CRETE, BSc nursing, Principal Investigator — Assistance Public-Hôpitaux de Paris; Medhi OUALHA, MD, PhD, Study Chair — Assistance Public-Hôpitaux de Paris
Locations (1):
- Necker Enfants malades hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebet RM, Hasbani NR, Sisko MT, Agus MSD, Nadkarni VM, Wypij D, Curley MAQ. Nurses' Perceptions of Workload Burden in Pediatric Critical Care. Am J Crit Care. 2021 Jan 1;30(1):27-35. doi: 10.4037/ajcc2021725. PMID 33385203
- [Background] Helmreich RL. On error management: lessons from aviation. BMJ. 2000 Mar 18;320(7237):781-5. doi: 10.1136/bmj.320.7237.781. No abstract available. PMID 10720367
- [Background] Llenore E, Ogle KR. Nurse-patient communication in the intensive care unit: a review of the literature. Aust Crit Care. 1999 Dec;12(4):142-5. doi: 10.1016/s1036-7314(99)70599-0. PMID 11271028
- [Background] Gurses AP, Carayon P, Wall M. Impact of performance obstacles on intensive care nurses' workload, perceived quality and safety of care, and quality of working life. Health Serv Res. 2009 Apr;44(2 Pt 1):422-43. doi: 10.1111/j.1475-6773.2008.00934.x. Epub 2008 Dec 16. PMID 19207589
- [Background] Nasirizad Moghadam K, Chehrzad MM, Reza Masouleh S, Maleki M, Mardani A, Atharyan S, Harding C. Nursing physical workload and mental workload in intensive care units: Are they related? Nurs Open. 2021 Jul;8(4):1625-1633. doi: 10.1002/nop2.785. Epub 2021 Feb 17. PMID 33596333
- [Background] Young G, Zavelina L, Hooper V. Assessment of workload using NASA Task Load Index in perianesthesia nursing. J Perianesth Nurs. 2008 Apr;23(2):102-10. doi: 10.1016/j.jopan.2008.01.008. PMID 18362006
- [Background] Tubbs-Cooley HL, Mara CA, Carle AC, Gurses AP. The NASA Task Load Index as a measure of overall workload among neonatal, paediatric and adult intensive care nurses. Intensive Crit Care Nurs. 2018 Jun;46:64-69. doi: 10.1016/j.iccn.2018.01.004. Epub 2018 Feb 12. PMID 29449130